CLINICAL TRIAL: NCT00160732
Title: Allogenic Islet Cells (Human, U. of Chicago) Administered Via Intraportal Infusion; and Immunosuppressive Therapy
Brief Title: Allogenic Islet Cell Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12176A; BB-IND 11228
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Islet Cell Transplant; Human islet cell infusion; Juvenile-onset diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplant (Experimental)
  Interventions: Drug: Allogenic islet cells (human, U. Chicago); Procedure: Intraportal infusion of islet cells

INTERVENTIONS:
Drug: Allogenic islet cells (human, U. Chicago) — Human allogenic islet cells. Immunosuppression varies but may include prograf, celcept, sirolimus, prednisone. Dosage will vary per patient based on weight. Patients will receive immunosuppression medications while islet cells are functioning.
Procedure: Intraportal infusion of islet cells — Intraportal infusion of islet cell through the portal vein in the liver.

SUMMARY:
The purpose of this study is to determine the safety of transplanting human islet cells for controlling hyperglycemia in brittle and/or complex patients with type 1 diabetes. In addition, initial observations will be made with regards to the effectiveness of reversing hypoglycemia with this treatment. The "Edmonton Protocol" of using specific anti-rejection drugs without steroids is also being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have type I diabetes mellitus, documented by undetectable C-peptide. Patients must have been diabetic for at least five years, and be aged 18 - 58 years.
* Patients must be on an intensive regimen of glucose monitoring and exogenous insulin injection (defined as greater than or equal to three checks and injections per day). This regimen must be prescribed and supervised by the patient's diabetologist.
* Despite intensive therapy, patients must have at least one of the following:

  * Brittle diabetes (metabolic instability), as defined by elevated mean amplitude of glycemic excursion;
  * Hypoglycemic unawareness, with at least one episode in the past two years in which hypoglycemia required the assistance of another person (e.g., family member, emergency medical technician [EMT], etc.), and was associated with a fingerstick blood glucose (FSBG) of < 50 mg/dl and prompt recovery after administration of oral glucose, intravenous glucose, or glucagon;
  * Progressive complications of diabetes (nephropathy manifested by proteinuria, retinopathy documented by an ophthalmologist after dilated eye exam, or neuropathy as determined by a neurologist).
* Patients must be able to give informed consent.

Exclusion Criteria:

* Failure to meet inclusion criteria
* Panel of Reactive Antibody (PRA) > 10%
* Creatinine clearance < 80 mL/min
* Prior organ transplant
* Portal hypertension: this refers to portal hypertension diagnosed previously by any means, or, by the investigators' evaluation, symptoms and/or signs of liver dysfunction with or without portal hypertension including, but not limited to, jaundice, ascites, encephalopathy, spider angiomata, coagulopathy, or peri-umbilical venous engorgement. Elevated portal pressures, as measured during intended islet infusion, may also result in discontinuation of infusion.
* Abnormal liver function tests (> 2 times the upper limit of normal as defined by the University of Chicago Clinical Laboratory)
* History of malignancy. Any history of malignancy in a patient who has had an "adequate" period of no evidence of neoplastic disease should not rule out individuals from enrolling in this study. Rather, pre-enrollment screening for malignancy will follow current established guidelines as for solid-organ transplant. These current guidelines appear in Kasiske, B.L., et al. "The Evaluation of Renal Transplant Candidates: Clinical Practice Guidelines," American Journal of Transplantation 1 (Supplement 2): 12-22, 2001.
* Active peptic ulcer disease
* Pregnancy, or inability to comply with contraceptive regimen
* Severe unremitting gastroparesis or diarrhea
* Active infection
* Serologic positivity for HIV and/or hepatitis
* Chest radiographic abnormality consistent with neoplastic or infectious disease
* Major ongoing psychiatric illness and/or substance abuse
* Noncompliance with current medical regimen
* Obesity (body mass index [BMI] > 28)
* Any other medical condition precluding safe transplantation and immunosuppression
* Ejection fraction < 30%
* Myocardial infarction (MI) within the past 6 months
* Known allergies or hypersensitivity to immunosuppressive agents used in this protocol
* Inability to provide written informed consent.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-10 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
decrease in insulin requirement - Subjects able to maintain fasting blood glucose concentrations below 126 mg/dL and 2-hour post prandial levels below 180 mg/dL will be considered to be insulin independent. | Monthly
decrease in incidence of hypoglycemic events | Monthly

SECONDARY OUTCOMES:
absence of complications from the procedure and side effects of the medication | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Witkowski, MD, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Hospitals, Chicago, Illinois, United States

REFERENCES:
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004